CLINICAL TRIAL: NCT03737149
Title: A Prospective Multicenter Longitudinal Cohort Study of the Mymobility Platform
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CLU2018-13CH
Record Dates: First submitted 2018-10-26; First posted 2018-11-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Knee Replacement; Knee Arthroplasty; Hip Replacement; Hip Arthroplasty; Joint Replacement; Physical Therapy; Partial Knee Replacement; Hip Pain, Chronic; Knee Pain, Chronic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: This is a staged cohort study. In the first (pilot) cohort, all participating subjects will utilize the mymobility with Apple Watch platform. In the second (RCT) cohort, approximately 1,000 subjects will be randomized 1:1 to either the mymobility with Apple Watch platform or standard of care SOC. In the third (correlative analytics) cohort, all participating subjects will utilize the mymobility with Apple Watch platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mymobility with Apple Watch (Experimental): Post-operative mobile application-guided education and exercise paired with accurate and sensitive activity monitoring.
  Interventions: Other: mymobility with Apple Watch
- Standard of Care Physical Therapy (No Intervention): Standard of care patient education and post-operative physical therapy, as determined by local site guidelines and care pathways.

INTERVENTIONS:
Other: mymobility with Apple Watch — The mymobility mobile application is a mobile software platform designed to facilitate remote episode of care management and asynchronous communication between the provider care team and their patient via provider-approved care plans and engagement communications. Current care pathways have been developed for: Total Hip Replacement, Total Knee Replacement and Partial Knee Replacement. Designed for the orthopedic population, mymobility also integrates wearable data from the Apple Watch into provider dashboards, providing enhanced understanding and monitoring of patients throughout the episode of care.
  Arms: mymobility with Apple Watch

SUMMARY:
Post-market prospective, multi-center longitudinal study to determine if mobile application-guided education and exercise paired with accurate and sensitive activity monitoring, captured from consumer wearables, can provide a viable (and potentially improved) alternative to current standard of care physical therapy for hip and knee arthroplasty.

DETAILED DESCRIPTION:
This is a post-market prospective, multi-center longitudinal study in subjects undergoing primary total knee arthroplasty (TKA), total hip arthroplasty (THA), or partial knee arthroplasty (PKA). The study objective is to determine if mobile application-guided education and exercise paired with accurate and sensitive activity monitoring, captured from consumer wearables, can provide a viable (and potentially improved) alternative to current standard of care patient education and physical therapy for hip and knee arthroplasty. The study will be conducted in phases. The first phase (N = 300) will consist of a pilot cohort of subjects and will primarily serve to determine site study staffing needs and time required for various elements of study execution. The second phase (N = 1,000, RCT) will consist of a randomized controlled subject cohort and will compare outcomes of mobile application-guided exercises and activity with standard of care (SOC) physical therapy. The third phase (N ~ 10,000 including subjects from both Phase I and the study arm from RCT/Phase II) will seek to collect enough data to enable the creation of decision support algorithms for outcomes of joint replacement. All subjects will undergo a TKA, THA, or PKA using SOC procedures and commercially-available devices as part of their clinical care. Subjects will then complete prescribed post-operative activities, such as physical therapy, according to SOC or performing exercises as scheduled through the mymobility app. In office assessments will be conducted at approximately 30 days prior to surgery, 30 days after surgery, and 3 months after surgery. Virtual assessments (including subject questionnaires and recording of adverse events) will occur at approximately 6 months and 1 year post-op.

February 2022 update: Eligibility criteria for new patients includes total knee and partial knee arthroplasty surgeries. Previously enrolled total hip arthroplasty patients will remain in the study for follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Subject must be 18 years of age or older.
2. Subject qualifies for a primary, unilateral total or partial knee arthroplasty, based on physical exam and medical history.
3. Investigator plans to treat subject with a commercially-available device, used on-label according to the manufacturer's instructions for use, as part of their clinical care.
4. Subject owns and maintains an iPhone capable of pairing to the Apple Watch, supporting iOS updates and is compatible with the mymobility App.
5. Subject is willing and able to complete the protocol required follow-up.
6. Subject is able to read and understand the language used in the mymobility App for their region.
7. Subject is willing and able to provide written Informed Consent and Authorization by signing and dating the IRB/EC approved Informed Consent Form and Authorization. Where applicable, subject must also be willing to provide authorization for use of protected health information in accordance with local privacy laws.
8. Subject is mobile with no more than a single cane/single crutch assist preoperatively.

Exclusion Criteria

1. Subject is a current alcohol or drug abuser as defined by the investigator.
2. Subject is considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.).
3. Subject has systemic inflammatory arthropathies which would interfere or compromise the activity profiles within this study.
4. Subject is currently participating in any other surgical intervention, physical therapy or pain management study which would compromise the results of this study.
5. Subject requires simultaneous or staged bilateral replacements, staged<90 days apart. Subjects can be enrolled into the study for the second, staged arthroplasty if scheduled >89 days after their first, contralateral replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10500 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase II (RCT): Readmission Rate | 30 Days postop
  RCT Phase: Non-inferiority of the mymobility with Apple Watch group in the number of readmissions through 30 days post-op compared to subjects receiving standard physical therapy.

SECONDARY OUTCOMES:
Phase II RCT: Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS, JR) | 90 Days
  The KOOS, JR score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Phase II RCT: Hip disability and Osteoarthritis Outcome Score - Joint Replacement (HOOS, JR) | 90 Days
  The HOOS, JR score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Phase II RCT: EQ-5D-5L | 90 Days
  Non-inferiority in post-operative EQ-5D-5L outcomes for the mymobility with Apple Watch group compared to subjects receiving standard physical therapy.
Phase II RCT: Incidence of Manipulation under Anesthesia (MUA) | 90 Days
  Comparison of incidence of Manipulation under anesthesia (MUA) between the study groups.
Phase II RCT: Timed Up and Go (TUG) | 90 Days
  Timed Up and Go Test: The time to rise from a chair, walk 10 feet, turn around, walk back to the chair and sit down.
Phase II RCT: Single-Leg Stance (SLS) Test | 90 Days
  Balance Test while standing on a single leg. Three tests are performed and the best of the three times is recorded. The maximum time for this test is 60 seconds.
Phase II RCT: Subject Satisfaction | 90 Days
  Comparison of subject satisfaction survey results between the study groups.
Phase II RCT: Healthcare Costs | 90 Days
  The number of hospital readmissions, reoperations, urgent care visits, and emergency room visits will be captured and used to calculate the cost of care after the joint replacement procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (30):
- United States (26):
  - Sah Orthopaedic Associates, Fremont, California
  - Hoag Orthopedic Institute, Irvine, California
  - Stanford University, Redwood City, California
  - Colorado Joint Replacement, Denver, Colorado
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Foundation for Orthopedic Research and Education, Temple Terrace, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Center for Joint Replacement, Indianapolis, Indiana
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - OrthoBethesda, Bethesda, Maryland
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Ascension Medical Group - University Orthopaedic Specialists, Rochester Hills, Michigan
  - Michigan Orthopaedic Surgeons, Troy, Michigan
  - Washington University, St Louis, Missouri
  - Rothman Institute, Montvale, New Jersey
  - New Mexico Orthopaedic Associates, Albuquerque, New Mexico
  - Duke University, Morrisville, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - JIS Orthopedics, New Albany, Ohio
  - Orthopedic + Fracture Specialists, Portland, Oregon
  - ROC Orthopedics, Tualatin, Oregon
  - Rothman Institute, Bryn Mawr, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - National Capital Private Hospital, Canberra, Australian Capital Territory
  - Epworth Healthcare - Richmond, Richmond, Victoria
- Policlinico Universitario Campus Bio-Medico, Roma, Italy
- St. Annaziekenhuis, Geldrop, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander JS, Redfern RE, Duwelius PJ, Berend KR, Lombardi AV Jr, Crawford DA. Use of a Smartphone-Based Care Platform After Primary Partial and Total Knee Arthroplasty: 1-Year Follow-Up of a Prospective Randomized Controlled Trial. J Arthroplasty. 2023 Jul;38(7 Suppl 2):S208-S214. doi: 10.1016/j.arth.2023.02.082. Epub 2023 Mar 6. PMID 36889524